CLINICAL TRIAL: NCT06597838
Title: Development and Validation of a Real-time Prediction Model for Acute Kidney Injury in Hospitalized Patients
Status: Recruiting | Type: Observational
Sponsor: Peking University First Hospital (Other)
Responsible Party: Principal Investigator, Li Yang, Professor, Peking University First Hospital
Other Study IDs: 2023[069-001]
Record Dates: First submitted 2024-09-09; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Prediction Model

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Early prediction of acute kidney injury (AKI) may provide a crucial opportunity for AKI prevention. To date, no prediction model targeting AKI among general hospitalized patients in developing countries has been published. We developed a simple, real-time, interpretable AKI prediction model for general hospitalized patients from a large tertiary hospital in China, and validated it across five independent, geographically distinct, different tiered hospitals.

DETAILED DESCRIPTION:
Early prediction of acute kidney injury (AKI) may provide a crucial opportunity for AKI prevention. To date, no prediction model targeting AKI among general hospitalized patients in developing countries has been published. We developed a simple, real-time, interpretable AKI prediction model for general hospitalized patients from a large tertiary hospital in China using the machine learning technique, and then validated the performance of the prediction model across five independent, geographically distinct, different tiered hospitals in China.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (18 years and older) admitted to five hospitals during the study period

Exclusion Criteria:

* Have less than 2 documented serum creatinine (Scr) measurements during hospitalization
* Being diagnosed with end-stage renal disease (ESRD)
* Maintained on dialysis or had an initial Scr greater than or equal to 4.0 mg/dL at admission
* Developed AKI prior to admission or within 24 hours after admission
* Length of stay shorter than 24 hours
* Underwent kidney transplantation or nephrectomy during hospitalization
* With all Scr measurements lower than or equal to 0.6 mg/dL from 90 days prior to admission until discharge.

Ages: 18 Years to 100 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult patients admitted to five hospitals during the study period.
Sampling Method: Probability Sample
Enrollment: 161876 (Estimated)
Dates: Start 2023-02-28 (Actual); Primary Completion 2024-10-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Predictive performance of the prediction model for Acute Kidney Injury | through study completion, varied from one to three years in different validation cohorts.
  Evaluated using AUC

CONTACTS AND LOCATIONS:
Overall Officials: Li Yang, Study Director — Peking University First Hospital
Locations (1):
- Peking University First Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No